CLINICAL TRIAL: NCT05032885
Title: RANDOMIZED CLINICAL TRIAL OF PHYSIOTHERAPY IN COVID PATIENTS ON THEIR PHYSICAL CONDITIONING, ANXIETY LEVEL AND THEIR QUALITY OF LIFE
Brief Title: Early Physiotherapy in Covid Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Principal Investigator, Susana Arias Rivera, Principal Investigator, Hospital Universitario Getafe
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIm20758
Record Dates: First submitted 2021-09-01; First posted 2021-09-02 (Actual); Last update posted 2023-03-29 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Insufficiency; Anxiety State
MeSH Terms: conditions — Respiratory Insufficiency; Anxiety Disorders | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (Experimental): 48-72 hours after hospital admission, following the baseline assessment of the patient, they will begin to receive physiotherapy treatment with respiratory techniques and motor training, adapted at all times to the clinical situation of the patient, until hospital discharge. If the patient's clinical condition worsens, treatment will be temporarily suspended until the patient improves to allow resumption of treatment.
  Interventions: Other: physiotherapy
- B (No Intervention): 48-72 hours after admission to the hospital, after the patient's baseline assessment, the patient will not receive physiotherapy and the usual referral to the Rehabilitation Service for physiotherapy treatment of hospitalized patients will be followed, if the patient's physician considers it necessary and requests it.

INTERVENTIONS:
Other: physiotherapy — Patients in the intervention group will receive early physiotherapy treatment. This intervention will consist of exercises and physiotherapy techniques commonly used and aimed at improving the patient's respiratory and motor conditioning.
  At the respiratory level: diaphragmatic and costal targeted ventilation, pursed-lip breathing and bronchial hygiene techniques if required.
  At the motor level: passive, active-assisted kinesitherapy and analytical and global potentiation of the upper and lower limbs that will allow the maintenance and improvement of the articular pathway and will prevent muscle weakness; retraining of transfers and balance; gait reeducation.
  Arms: A

SUMMARY:
Based on the hypothesis that early physiotherapy in patients hospitalized for COVID-19 improves their functional capacity, perceived quality of life and decreases anxiety. Our main objective is to analyze the differences between groups with respect to functional deterioration, need for oxygen therapy and anxiety when implementing an early physiotherapy program.

We propose a randomized clinical trial with two arms and single-center, to be developed in hospitalization units and intermediate respiratory care units (IRCU), with patients diagnosed with COVID. The sample will consist of an experimental group of 66 admitted patients with COVID-19 to whom an early physiotherapy program will be implemented from 48-72 hours after admission. The control group will be made up of another 66 admitted patients with COVID-19 who will receive the treatment according to the usual procedure of the hospital center.

Sociodemographic and clinical variables will be collected, including: modified MMRC dyspnea scale, amount of oxygen therapy, MRC-SS, sit to stand test, hand grip, Tinetti, HADS anxiety and depression questionnaire, SF-12 quality of life questionnaire, clinical frailty scale (CFS) and FRAIL scale. Patients in both groups will be re-evaluated two months after hospital discharge with the above variables in addition to the PCFS post-COVID patient functional status scale.

A basic descriptive analysis and logistic regression will be performed to determine the effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the hospitalization unit or intermediate respiratory care unit, diagnosed with COVID-19 pneumonia, of legal age and who consent to participate in the study. Pregnant patients or patients with dementia, terminal illnesses or those in which there are communication problems (language problems, comprehension ...) will not be included.

Exclusion Criteria:

* Patients who are transferred to another acute hospital due to impossibility of completing the follow-up period, exitus during hospital admission and those who revoke consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2021-04-04 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Respiratory competence | 4 months
  Monitoring and assessment of the respiratory capacity of patients during hospital admission
Motor competence | 4 months
  Monitoring and assessment of patients' motor skills during hospital admission

SECONDARY OUTCOMES:
Anxiety state | 4 months
  assessment of the anxiety state of patients on admission and after discharge from hospital
Variation in the level of quality of life | 4 months
  Assessment of patients' quality of life prior to hospital admission and two months after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Susana Arias-Rivera, Getafe, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No